CLINICAL TRIAL: NCT05902728
Title: Study on Food Influence and Drug-drug Interaction of HLX208 Tablets in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-PK-001
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: NSCLC
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX208 in the fast state (Experimental): HLX208 900mg in the fast state
  Interventions: Drug: HLX208
- HLX208 in the fed state (Experimental): HLX208 900mg in the fed state
  Interventions: Drug: HLX208
- HLX208 + Itraconazole group (Experimental): HLX208 + Itraconazole group
  Interventions: Drug: HLX208; Drug: Itraconazole 200 mg
- HLX208 + rifampicin group (Experimental): HLX208 + rifampicin group
  Interventions: Drug: HLX208; Drug: Rifampicin

INTERVENTIONS:
Drug: HLX208 — Subjects will receive treatment HLX208 900 mg in the fast state followed by 7 days washout ，then receive treatment HLX208 900 mg in the fed state
  Arms: HLX208 in the fast state
Drug: HLX208 — Subjects will receive treatment HLX208 900 mg in the fed state followed by 7 days washout ，then receive treatment HLX208 900 mg in the fast state.
  Arms: HLX208 in the fed state
Drug: HLX208 — 450 mg
  Arms: HLX208 + Itraconazole group
Drug: HLX208 — 900 mg
  Arms: HLX208 + rifampicin group
Drug: Itraconazole 200 mg — 200 mg
  Arms: HLX208 + Itraconazole group
Drug: Rifampicin — 600mg
  Arms: HLX208 + rifampicin group

SUMMARY:
This study is divided into Part I and Part II. Part I is the food effect study. A total of 20 healthy subjects, regardless of gender, will be enrolled in a randomized, open-label, crossover design.

Part II is the drug-drug interaction study, an open-label and sequential design. 32 healthy subjects are planned to be enrolled and divided into group A and group B. Group A is to evaluate the influence of itraconazole as CYP3A4 strong inhibitory on HLX208. Group B was to evaluate the effect of rifampicin as a strong inducer of CYP3A4 on HLX208.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the content, process and possible adverse reactions of the trial. Must be able to communicate with the investigator, understand and comply with all study requirements;
2. Male or female subjects aged 18 to 45 (including 18 and 45);
3. Weigh at least 50 kg (for male) and 45 kg (for female), respectively, and have a body mass index (BMI) ≥ 19 and ≤26 kg/m2. BMI = weight (kg)/[height (m)]2;

Exclusion Criteria:

1. Known history of drug or food allergy;
2. Those who have a positive urine drug screen or have a history of drug abuse;
3. Excessive smoking (≥ 5 cigarettes/day);

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter Cmax of HLX208 | up to 48 hours
  Cmax of HLX208
Pharmacokinetics parameter AUC0-t of HLX208 | up to 48 hours
  AUC0-t of HLX208
Pharmacokinetics parameter AUC0-inf of HLX208 | up to 48 hours
  AUC0-inf of HLX208

SECONDARY OUTCOMES:
other pharmacokinetics parameter Tmax of HLX208 | up to 48 hours
  Tmax of HLX208
other pharmacokinetics parameter Tlag of HLX208 | up to 48 hours
  Tlag of HLX208
other pharmacokinetics parameter t1/2 of HLX208 | up to 48 hours
  t1/2 of HLX208
other pharmacokinetics parameter CL/F of HLX208 | up to 48 hours
  CL/F of HLX208
other pharmacokinetics parameter Vd/F of HLX208 | up to 48 hours
  Vd/F of HLX208
other pharmacokinetics parameter MRT of HLX208 | up to 48 hours
  MRT of HLX208
other pharmacokinetics parameter %AUCex of HLX208 | up to 48 hours
  %AUCex of HLX208
The incidence and severity of adverse events/serious adverse events | up to 17 days after the last dose
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No